CLINICAL TRIAL: NCT06975540
Title: Study of the Synergy Between Physical Exercise and a Nutritional Supplement for the Prevention and Treatment of Frailty: The ROBUSTNES Study
Brief Title: Synergy of Exercise and Nutrition in Preventing and Treating Frailty
Acronym: ROBUSTNES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: University of Valencia (Other); Nestle Health Science (Industry); Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Principal Investigator, Maria Carmen Gómez Cabrera, PhD, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEJ-NES-2019; PID2019-110906RB-100 (Other Grant/Funding Number: Ministry of Science of Spain); MEJ-NES-2019 (Other Grant/Funding Number: Nestlé Health Sicence S.A.)
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Frail Elderly
Keywords: Frailty; Malnutrition; Physical exercise program; Nutritional supplementation
MeSH Terms: conditions — Frailty; Malnutrition

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants take the nutritional supplement (MERITENE, 30g twice a day) and attend supervised exercise sessions as part of the multicomponent program (3days/week) for 180 days.
  Interventions: Other: Multidomain physical exercise
- Control (No Intervention): Participants receive neither.

INTERVENTIONS:
Other: Multidomain physical exercise — The intervention includes a daily intake of two 200-mL of Meritene nutritional supplements (199 Kcal, 16g of protein, 25g of carbs, 3.6g of fats, and enriched with vitamins and minerals/bottle) plus a supervised and personalized multicomponent exercise program. Multicomponent exercise program (MEP) includes endurance, strength, coordination, balance, and flexibility exercises. The sessions last 65 min a day, 3 days/week for 24 weeks. All the sessions are supervised and delivered in groups by sports scientists.
  Arms: Intervention

SUMMARY:
The goal of this clinical study is to learn if combining a nutritional supplement with a multicomponent exercise program can help prevent and treat frailty in community dwelling older adults. The main questions it aims to answer is: Does combining a nutritional supplement (MERITENE) with a multicomponent exercise program improve frailty and functionality in older adults?

Researchers will compare:

* A group receiving both the nutritional supplement and the exercise program (intervention group)
* A control group receiving neither (control group)

Participants:

* take the nutritional supplement (MERITENE, 30g twice a day) for 180 days
* attend (3days/week) supervised exercise sessions as part of the multicomponent program for 180 days (if assigned to the intervention group).
* undergo regular clinical evaluations for frailty, nutritional status, cognitive function, emotional state, and quality of life.

Measurements will include: Changes in frailty status, particularly gait speed, measured using Share-fi criteria, nutritional assessment using the Mini Nutritional Assessment (MNA), physical and cognitive assessments, including Edmonton Frail Scale, MMSE, and Short Physical Performance Battery (SPPB) and a complete biochemical and clinical blood analysis.

ELIGIBILITY:
Inclusion Criteria:

* i) men and women aged 70 years or older; ii) sedentary (less than three hours of weekly physical activity), iii) frail according to the Survey of Health, Ageing and Retirement in Europe Frailty Index (SHARE-FI); iv) gait speed lower or equal than 0.8 m/sec, v) community dwellers

Exclusion Criteria:

* i) life expectancy from the moment of selection lower than twelve months by any cause; ii) poorly controlled diabetes (glycated hemoglobin > 9%); iii) cognitive impairment (score less than 17 in the MMSE); iv) disability (score less than 50 points on Barthel's Scale); v) acute coronary event in the previous year; vi) hospital admission in the previous three months for any reason; vii) oncologic patient with active treatment with chemotherapy or radiotherapy; viii) major non-ambulatory surgery in the previous six months; ix) patient with a coronary event in the previous twelve months; x) institutionalized patient; xi) New York Heart Association class 3 to 4 baseline dyspnea; xii) lactose intolerance; xiii) being supplemented with a multivitamin or a protein-rich food; xiv) refusal to sign the informed consent.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Frailty according to the Survey of Health, Ageing and Retirement in Europe Frailty Index (SHARE-FI) | 24 weeks (180 days)
  Change in frailty status assessed by Fried's criteria after 180 days.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia /Hospital Clínico Universitario de València, Valencia, Spain, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garcia-Gimenez JL, Mena-Molla S, Tarazona-Santabalbina FJ, Vina J, Gomez-Cabrera MC, Pallardo FV. Implementing Precision Medicine in Human Frailty through Epigenetic Biomarkers. Int J Environ Res Public Health. 2021 Feb 15;18(4):1883. doi: 10.3390/ijerph18041883. PMID 33672064
- [Background] Millan-Domingo F, Tarazona-Santabalbina FJ, Carretero A, Olaso-Gonzalez G, Vina J, Gomez-Cabrera MC. Real-Life Outcomes of a Multicomponent Exercise Intervention in Community-Dwelling Frail Older Adults and Its Association with Nutritional-Related Factors. Nutrients. 2022 Dec 3;14(23):5147. doi: 10.3390/nu14235147. PMID 36501177
- [Background] Arc-Chagnaud C, Millan F, Salvador-Pascual A, Correas AG, Olaso-Gonzalez G, De la Rosa A, Carretero A, Gomez-Cabrera MC, Vina J. Reversal of age-associated frailty by controlled physical exercise: The pre-clinical and clinical evidences. Sports Med Health Sci. 2019 Sep 10;1(1):33-39. doi: 10.1016/j.smhs.2019.08.007. eCollection 2019 Dec. PMID 35782461